CLINICAL TRIAL: NCT05819853
Title: Role of Semaglutide in Restoring Ovulation in Youth and Adults With Polycystic Ovary Syndrome
Acronym: RESTORE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-4941; R01HD108340 (NIH)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; Obese
Keywords: PCOS; semaglutide
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Untreated PCOS (Experimental): Participants with PCOS who are not on metformin or hormonal therapy, will receive 10-months of semaglutide intervention.
  Participants will get either semaglutide as either:
  Wegovy: 0.25mg for 4 weeks, 0.5mg for 4 weeks, 1mg 4-weeks, and 1.7mg for the remainder of the study.
  or
  Ozempic: 0.25mg for 4 weeks, 0.5mg for 4 weeks, 1mg 4-weeks, and Wegovy for 1.7mg for the remainder of the study.
  Interventions: Drug: Semaglutide Injectable Product (Wegovy and/or Ozempic)
- PCOS on Metformin (Experimental): Participants with PCOS who are currently on metformin and still not having regular menses, will receive 10-months of semaglutide intervention. Participants in this arm will continue to take their metformin throughout the trial.
  Participants will get either semaglutide as either:
  Wegovy: 0.25mg for 4 weeks, 0.5mg for 4 weeks, 1mg 4-weeks, and 1.7mg for the remainder of the study.
  or
  Ozempic: 0.25mg for 4 weeks, 0.5mg for 4 weeks, 1mg 4-weeks, and Wegovy for 1.7mg for the remainder of the study.
  Interventions: Drug: Semaglutide Injectable Product (Wegovy and/or Ozempic)

INTERVENTIONS:
Drug: Semaglutide Injectable Product (Wegovy and/or Ozempic) — 10 months of semaglutide, with dose escalation as recommended by manufacturer. Maximum dose used will be 1.7mg
  Other Names: Semaglutide (Wegovy and/or Ozempic)

SUMMARY:
Girls and women 12-35 years old with obesity and polycystic ovarian syndrome who are on or off metformin, will receive a glucagon like peptide-1 receptor agonist intervention for 10 months to induce metabolic changes, weight loss and improve reproductive abnormalities.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is one of the most common endocrinopathies in women, presents with anovulation in adolescence, and reproductive dysfunction is related to excess weight. After a 4-month observation period of either no medication or metformin treatment, females aged 12-35 years with obesity and polycystic ovary syndrome will receive 10 months of a glucagon-like peptide-1 receptor agonist to induce metabolic changes, weight loss and improve reproductive abnormalities. We will assess the relationship between weight loss and reproductive function, as well as identify if age, hormonal and metabolic measures and such insulin sensitivity and insulin secretion predict the response to glucagon-like peptide-1 receptor agonist therapy.

ELIGIBILITY:
Inclusion Criteria

1. Female
2. Ages 12-35 years
3. Sedentary- less than 2 hours of moderate (jogging, swimming etc.) exercise a week.
4. Oligomenorrhea, on or off metformin, as defined per age category in the most recent 2018 PCOS international guidelines
5. Initial BMI based on age and weight:

   1. If <18 years, initial BMI percentile ≥95
   2. If 18-35 years, initial BMI ≥30 kg/m2 OR initial BMI ≥27 kg/m2 with at least one weight-related comorbid condition, e.g., hypertension or dyslipidemia
   3. Must be weight stable within ±5kg in the 3 months prior to enrollment
6. Diagnosed with PCOS per the most stringent NIH criteria with adaptation for adolescents (oligomenorrhea >24 months post-menarche or primary amenorrhea after age 15 years and clinical/ biochemical hypertestosteronemia
7. Participants cannot be on hormonal contraception, so participants should remain abstinent or use reliable non-hormonal contraception (e.g., copper IUD) for the entire study period. For participants who receive semaglutide, they should avoid pregnancy for at least 2 months after stopping medication to avoid fetal exposure to the medication.
8. For participants in the metformin + semaglutide group, participants must have been stable on ≥ 1500 mg of metformin a day for at least 3 months by time of screening

Exclusion Criteria:

1. Diagnosed with or have a family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN2). Family history of medullary thyroid cancer or thyroid nodule palpated by endocrinologist at screening. - Per approved drug label
2. Use of medications known to affect insulin sensitivity: metformin (cannot have been used in the 3 months prior to screening for the untreated arm of the study), chronic oral steroids, oral glucocorticoids within 10 days, atypical antipsychotics, immunosuppressant agents, HIV medications, estrogen-containing hormonal contraception (cannot have been used in the 6 months prior to screening), progesterone-containing hormonal contraception (cannot have been used in the 3 months prior to screening). Dermal patch or vaginal ring contraception methods. Weight loss medications or stimulants. Use of other products containing other GLP-1 agonists.
3. Weight loss medications in the last 6 months
4. Currently pregnant or breastfeeding women. Development of pregnancy during the study period will necessitate withdrawal from the study.
5. Severe illness requiring hospitalization within 60 days.
6. Diabetes, defined as Hemoglobin A1C ≥6.5%
7. Anemia, defined as Hemoglobin < 12 mg/dL
8. Diagnosed major psychiatric or developmental disorder limiting informed consent.

10) Known liver disease other than NAFLD, or AST or ALT >125 IU/L. 11) Personal history of pancreatitis 12) Known renal disease of any severity or an eGFR at screening of <45ml/min/1.73m2 13) History of severe GI disease (e.g., gastroparesis) 14) History of gallstones 15) Untreated thyroid disease 16) History of hypersensitivity to semaglutide 17) Other causes of hyperandrogenism (example: tumor, CAH) or amenorrhea (untreated thyroid disease, tumor, primary ovarian failure, prolactinoma).

18) Active symptoms or undergoing treatment for anorexia nervosa or binging/purging disorder 19) Desiring pregnancy in the next 12-18 months. 20) Bariatric surgery 21) Use of THC (smoking or edible) more than 3 days a week 22) Alcohol use-drinking more than 2 drinks, more than 3 days a week 23) Any potential participants who cannot/will not commit to abstinence, use of a copper intrauterine device (IUD), or use of double barrier forms of contraception.

Ages: 12 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — PCOS is a condition only found in those of female sex
Enrollment: 80 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in ovulation frequency before and after semaglutide in females with PCOS | 14 months
  The change in ovulation will be measured at baseline and 6-10 months post treatment with semaglutide from 4 months daily urinary progesterone metabolites

SECONDARY OUTCOMES:
Change in Whole Body Insulin Sensitivity | Baseline and 10 months
  Participants will undergo a 75 gram oral glucose tolerance test, and whole body insulin sensitivity will be expressed as Si, calculated via the oral minimal model using SAMM II software. This software uses participant weight, glucose and insulin concentrations at various time points during the oral glucose tolerance test to calculate the participant's insulin sensitivity. A positive Si value means an improvement in insulin sensitivity.
Change in ovarian morphology | Baseline and 10 months
  Participants will have an ovarian ultrasound performed to measure change in ovarian morphology: ovarian size and number of follicles pre/post treatment with semaglutide

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Cree-Green, MD,PhD, Principal Investigator — University of Colorado Anschutz/Children's Hospital Colorado
Locations (1):
- University of Colorado Anschutz/Children's Hospital Colorado Aurora, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No